CLINICAL TRIAL: NCT03581227
Title: The CAPTURE Study: Validating a Unique Chronic Obstructive Pulmonary Disease (COPD) Case Finding Tool in Primary Care
Brief Title: The CAPTURE Study: Validating a Unique COPD Case Finding Tool in Primary Care (Aim 1)
Acronym: CAPTURE
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); University of Michigan (Other); National Jewish Health (Other); University of Minnesota (Other); Duke University (Other); Wake Forest University Health Sciences (Other); Oregon Health and Science University (Other); High Plains Research Network (Network); L.A. Net Community Health Resource Network (Other); COPD Foundation (Other); University of Kentucky (Other)
Responsible Party: Sponsor
Other Study IDs: 1803019032-1; R01HL136682-01 (NIH)
Record Dates: First submitted 2018-06-26; First posted 2018-07-10 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: CAPTURE, COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants without a diagnosis of COPD: Men and women aged 45 to 80, who have not been diagnosed with Chronic Obstructive Pulmonary Disease (COPD)
  Interventions: Other: CAPTURE Tool

INTERVENTIONS:
Other: CAPTURE Tool — CAPTURE Tool: a self administered 5-item questionnaire with peak expiratory flow measurements

SUMMARY:
A prospective multi-center study to define the sensitivity and specificity of CAPTURE for identifying previously undiagnosed patients with clinically significant COPD in a broad range of primary care settings.

DETAILED DESCRIPTION:
The CAPTURE tool consists of a 5-item self-administered questionnaire and selected use of peak expiratory flow (PEF) measurement, designed to identify clinically significant COPD.

For Aim 1 approximately 5,000 patients will be recruited across 100 participating primary care clinics. Eligible participants will undergo a baseline visit during which the CAPTURE tool and PEF will be obtained, as well as spirometry and other participant characteristics.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, aged 45-80 years

Exclusion Criteria:

1. Previous clinician provided diagnosis of COPD
2. Treated respiratory infection (with antibiotics and/or systemic steroids) in the past 30 days of baseline
3. Participants unable to perform spirometry due to any of the following conditions within the past 30 days of baseline

   1. Chest surgery
   2. Abdominal surgery
   3. Eye surgery
   4. Heart attack
   5. Stroke

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult men and women recruited from a broad range of primary care settings across the United States.
Sampling Method: Probability Sample
Enrollment: 4679 (Actual)
Dates: Start 2018-10-12 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of CAPTURE to identify previously undiagnosed patients with clinically significant COPD at baseline | Baseline
  Sensitivity and specificity of CAPTURE to identify previously undiagnosed patients with clinically significant COPD at baseline. Clinically significant COPD is defined as participants with abnormal spirometry, defined as post-bronchodilator FEV1/FVC < 0.7, plus one of the following: FEV1 < 60% predicted, or ≥ 1 exacerbation-like event within the past 12 months.
  If a participant is unable to complete a post-bronchodilator spirometry (refusal, technical error on the part of coordinator, etc.), and the pre-bronchodilator FEV1/FVC is less than 0.65, the participant will be considered to have COPD for the purpose of follow-up in this study.

SECONDARY OUTCOMES:
Sensitivity and specificity of CAPTURE to identify previously undiagnosed patients with clinically significant COPD across sex, ethnic groups, urban vs rural location, and educational status. | Baseline
  Sensitivity and specificity of CAPTURE to identify previously undiagnosed patients with COPD across sex, ethnic groups, urban vs rural location, and educational status.
Positive and negative predictive values (PPV and NPV) in different practice settings | Baseline
  Positive and negative predictive values in different practice settings
Areas under the receiving operator characteristic curve (AUC) for various cutpoints of CAPTURE and PEF (Peak expiratory flow) measurements to determine the best cutpoint for clinically significant COPD screen | Baseline
  AUC for various cutpoints of CAPTURE and PEF measurements to determine the best cutpoint for clinically significant COPD screen.
AUC to identify the combination of patient/site characteristics which best discriminates those with clinically significant COPD | Baseline
  AUC to identify the combination of patient/site characteristics which best discriminates those with clinically significant COPD
Sensitivity and specificity of CAPTURE to identify previously undiagnosed patients with spirometrically defined COPD at baseline | Baseline
  Sensitivity and specificity of CAPTURE to identify previously undiagnosed patients with Spirometrically defined COPD at baseline. Spirometrically defined COPD is defined as post-bronchodilator FEV1/FVC < 0.70.
Sensitivity and specificity of CAPTURE to identify previously undiagnosed patients with spirometrically defined COPD across sex, ethnic groups, urban vs rural location, and educational status. | Baseline
  Sensitivity and specificity of CAPTURE to identify previously undiagnosed patients with spirometrically defined COPD across sex, ethnic groups, urban vs rural location, and educational status. Spirometrically defined COPD is defined as post-bronchodilator FEV1/FVC < 0.70
Areas under the receiving operator characteristic curve (AUC) for various cutpoints of CAPTURE and PEF (Peak expiratory flow) measurements to determine the best cutpoint for spirometrically defined COPD screen | Baseline
  AUC for various cutpoints of CAPTURE and PEF measurements to determine the best cutpoint for spirometrically defined COPD (FEV1/FVC < 0.70) screen.
AUC to identify the combination of patient/site characteristics which best discriminates those with spirometrically defined COPD | Baseline
  AUC to identify the combination of patient/site characteristics which best discriminates those with spirometrically defined COPD (FEV1/FVC < 0.70).
Sensitivity and specificity of CAPTURE to identify previously undiagnosed patients with mild COPD at baseline | Baseline
  Sensitivity and specificity of CAPTURE to identify previously undiagnosed patients with mild COPD at baseline. Mild COPD is defined as participants with abnormal spirometry, defined as post-bronchodilator FEV1/FVC < 0.7, plus both of the following: FEV1 > 60% predicted and no prior history of COPD exacerbation.
Sensitivity and specificity of CAPTURE to identify previously undiagnosed patients with mild COPD across sex, ethnic groups, urban vs rural location, and educational status. | Baseline
  Sensitivity and specificity of CAPTURE to identify previously undiagnosed patients with mild COPD across sex, ethnic groups, urban vs rural location, and educational status. Mild COPD is defined as participants with abnormal spirometry, defined as post-bronchodilator FEV1/FVC < 0.7, plus both of the following: FEV1 > 60% predicted and no prior history of COPD exacerbation.
Areas under the receiving operator characteristic curve (AUC) for various cutpoints of CAPTURE and PEF (Peak expiratory flow) measurements to determine the best cutpoint for mild COPD screen | Baseline
  AUC for various cutpoints of CAPTURE and PEF measurements to determine the best cutpoint for mild COPD screen. Mild COPD is defined as participants with abnormal spirometry, defined as post-bronchodilator FEV1/FVC < 0.7, plus both of the following: FEV1 > 60% predicted and no prior history of COPD exacerbation.
AUC to identify the combination of patient/site characteristics which best discriminates those with mild COPD | Baseline
  AUC to identify the combination of patient/site characteristics which best discriminates those with mild COPD. Mild COPD is defined as participants with abnormal spirometry, defined as post-bronchodilator FEV1/FVC < 0.7, plus both of the following: FEV1 > 60% predicted and no prior history of COPD exacerbation.

CONTACTS AND LOCATIONS:
Overall Officials: Fernando J Martinez, MD, MS, Principal Investigator — Weill Medical College of Cornell University; MeiLan Han, Principal Investigator — University of Michigan
Locations (8):
- United States (8):
  - LANet, Los Angeles, California
  - High Plains Research Network, Aurora, Colorado
  - COPD Foundation, Miami, Florida
  - Cook County Health, Chicago, Illinois
  - University of Illinois at Chicago, Chicago, Illinois
  - Atrium Healthcare, Charlotte, North Carolina
  - Duke University, Durham, North Carolina
  - Oregon Rural Practice-based Research Network (ORPRN), Portland, Oregon

REFERENCES:
- [Derived] Martinez FJ, Yawn BP, Angulo D, Lopez C, Murray S, Mannino D, Anderson S, Dolor R, Elder N, Joo M, Khan I, Knox LM, Meldrum C, Peters E, Spino C, Tapp H, Thomashow B, Zittleman L, Brown R, Make B, Han MK; CAPTURE Study Group. Impact of the CAPTURE Chronic Obstructive Pulmonary Disease Screening Tool in U.S. Primary Care: A Cluster-Randomized Trial. Am J Respir Crit Care Med. 2025 May;211(5):789-802. doi: 10.1164/rccm.202405-0921OC. PMID 39715575